CLINICAL TRIAL: NCT04872023
Title: Immunomonitoring and Multiple Myeloma: Impact of Lenalidomide on Immune Checkpoint
Brief Title: Immunomonitoring and Multiple Myeloma: Impact of Lenalidomide on Immune Checkpoint Expression
Acronym: IMMUNO-MYELO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC17_8825_IMMUNOMYELO
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): All patients will have a extra blood sampling before first cycle of treatment and after one cycle. They also have an extra bone marrow sampling after the first cycle of treatment
  Interventions: Other: Blood and bone marrow sampling

INTERVENTIONS:
Other: Blood and bone marrow sampling — Blood and bone marrow sampling

SUMMARY:
The myeloma microenvironment is the target of many drugs in development, and it is unclear how they can be combined with reference treatments such as lenalidomide. This pilot study consists of an extensive phenotypic characterisation of the impact of lenalidomide combined with dexamethasone on the bone marrow microenvironment of a homogeneous cohort of non-pretreated MM patients. Blood sampling will be systematically performed in a matched fashion to monitor the general effect of lenalidomide on the immune system and to detect possible peripheral markers.

This study will provide rational guidance for future combination therapies with lenalidomide.

DETAILED DESCRIPTION:
With the significant increase in the number of therapeutic combinations targeting the tumour microenvironment, it is crucial to better understand the effect of reference myeloma treatments on the different immune populations present in the tumour in order to rationally optimise the combination with new strategies under development. In addition, the identification of biomarkers in the circulating blood that can predict/monitor the impact of new therapies on the immune response is a major challenge.

This pilot study consists of an extensive phenotypic characterisation of the impact of lenalidomide combined with dexamethasone on the bone marrow microenvironment of a homogeneous cohort of non-pretreated MM patients. Blood sampling will be systematically performed in a matched fashion to monitor the general effect of lenalidomide on the immune system and to detect possible peripheral markers.

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed multiple myeloma;
* Patient not eligible for intensive treatment;
* Patient for whom first-line treatment with Lenalidomide-Dexamethasone will be initiated;
* Patient accepting the performance of an additional myelogram at the end of the 1st treatment cycle.
* Patient aged 18 years or older;
* Patient who has given free, informed and written consent;
* Patient affiliated to a social security scheme
* For women of childbearing age, use of effective contraception

Exclusion Criteria:

* Patient with relapsed multiple myeloma;
* Patient eligible for intensive treatment;
* Patient for whom chemotherapy involves treatment other than Lenalidomide-Dexamethasone;
* Patient with a contraindication to lenalidomide treatment
* Pregnant or breastfeeding woman;
* Person subject to legal protection (safeguard of justice, curatorship,guardianship) or person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Rate of HLA-DR on medullary T-lymphocytes | 1 month
  Changed expression of HLA-DR on medullary T-lymphocytes after exposure to lenalidomide-dexamethasone.

SECONDARY OUTCOMES:
Activation status of biological markers | 1 month
  Presence of active protein markers and immune checkpoints by medullary immune cell subpopulations.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No